CLINICAL TRIAL: NCT00702377
Title: Evaluation of SYSTANE Ultra Lubricant Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-07-33
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2010-02-10 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SYSTANE Ultra (Experimental): SYSTANE Ultra Lubricant Eye Drops
  Interventions: Other: SYSTANE Ultra
- OPTIVE (Active Comparator): OPTIVE Lubricant Eye Drops
  Interventions: Other: Optive

INTERVENTIONS:
Other: SYSTANE Ultra — SYSTANE Ultra Lubricant Eye Drops 1 drop each eye 4 times daily for 42 days
  Arms: SYSTANE Ultra
Other: Optive — Optive Lubricant Eye Drops 1 drop each eye 4 times daily for 42 days
  Arms: OPTIVE

SUMMARY:
To evaluate the safety and efficacy of two artificial tears in dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of dry eyes
* Must not have worn contact lenses for 1 week preceding enrollment

Exclusion Criteria:

* Age related

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Call Center for Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 109 dry eye subjects
Pre-assignment Details: Randomized, double-masked, parallel design
Groups:
- OPTIVE Lubricant Eye Drops: OPTIVE Lubricant Eye Drops 1 drop each eye 4 times daily for 42 days
Period: Overall Study
Arm/Group | SYSTANE Ultra | OPTIVE Lubricant Eye Drops
Started | 53 | 56
Completed | 52 | 53
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SYSTANE Ultra | OPTIVE Lubricant Eye Drops | Total
Number analyzed (Participants) | 53 | 56 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 43 | 77
  >=65 years | 19 | 13 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 41 | 80
  Male | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Tear Break-up Time
Description: Tear breakup time is the time interval between a blink and the development of a dry spot in the tear film. Less than 10 seconds is abnormal. Dry spot is visible after fluorescein staining when viewed under a slit-lamp.
Time Frame: Day 0, Day 7, Day 14, Day 28, and Day 42
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | SYSTANE Ultra | OPTIVE Lubricant Eye Drops
Number analyzed (Participants) | 53 | 56
seconds
  Day 0 | 4.2 (1.9) | 4.5 (2.3)
  Day 7 | 4.7 (2.8) | 4.2 (1.8)
  Day 14 | 4.8 (2.8) | 4.2 (1.8)
  Day 28 | 4.6 (2.6) | 5.2 (3.2)
  Day 42 | 4.5 (2.3) | 4.2 (2.3)

2. Primary Outcome: Conjunctival Staining
Description: Conjunctival staining refers to the appearance of spots on the conjunctiva when dyed with lissamine green stain during an eye examination. Lissamine green temporarily stains the surface of the conjunctiva of the eye. An eye doctor looking at the eye's surface through a slit lamp observes the spots as green spots. Conjunctival staining grading scale is a 6 point scale, with 0 equals no staining (best case) and 6 equals maximum (worst) staining.
Time Frame: Day 0, Day 7, Day 14, Day 28, Day 42
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SYSTANE Ultra | OPTIVE Lubricant Eye Drops
Number analyzed (Participants) | 53 | 56
Units on a scale
  Day 0 | 2.3 (1.1) | 2.8 (1.4)
  Day 7 | 2.1 (1.1) | 2.5 (1.3)
  Day 14 | 2.0 (1.2) | 2.2 (1.4)
  Day 28 | 1.9 (1.1) | 2.4 (1.5)
  Day 42 | 1.9 (1.0) | 2.7 (1.4)

3. Primary Outcome: Corneal Staining
Description: Corneal staining refers to the appearance of corneal abrasions when dyed with fluorescein drops during an eye examination. Fluorescein temporarily stains the surface of the cornea of the eye. An eye doctor looking at the eye's surface through a slit lamp observes the abrasions as brightly-colored spots on an otherwise smooth cornea. Corneal staining grading scale is a 15 point scale, with 0 equals no staining (best case) and 15 equals maximum (worst) staining.
Time Frame: Day 0, Day 7, Day 14, Day 28, Day 42
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SYSTANE Ultra | OPTIVE Lubricant Eye Drops
Number analyzed (Participants) | 53 | 56
Units on a scale
  Day 0 | 4.8 (1.8) | 5.3 (2.5)
  Day 7 | 3.6 (2.2) | 4.3 (3.0)
  Day 14 | 2.9 (2.1) | 4.5 (2.9)
  Day 28 | 3.1 (2.1) | 3.8 (2.6)
  Day 42 | 2.9 (1.8) | 4.2 (2.8)

ADVERSE EVENTS:
Time Frame: From Day 0 to Day 42.
Description: Adverse events were both volunteered and solicited.
Arm/Group | SYSTANE Ultra | OPTIVE Lubricant Eye Drops
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/56
Other Adverse Events (participants affected / at risk) | 3/53 | 0/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYSTANE Ultra (N=53) | OPTIVE Lubricant Eye Drops (N=56)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI should hold confidential, and not disclose directly or indirectly to any third party other than Contractors, the data arising out of the study. Alcon reserves the right of prior review of any publication or presentation of information related to the study.